CLINICAL TRIAL: NCT02553772
Title: A Multicenter, Double-masked, Randomized Study to Compare the Safety and Efficacy of the OM3 Tear Formulation With REFRESH OPTIVE® ADVANCED Unit Dose for 3 Months in Patients With Dry Eye Disease
Brief Title: A Safety and Efficacy Study of a New Eye Drop Formulation in Patients With Dry Eye Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11182X-001
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OM3 Tear (Experimental): Carboxymethylcellulose based eye drop [Omega-3 (OM3) Tear] administered as 1-2 drops in each eye, as needed, at least 2 times daily for 90 days.
  Interventions: Drug: Carboxymethylcellulose Based Eye Drop
- REFRESH OPTIVE® ADVANCED (Active Comparator): Carboxymethylcellulose sodium 0.5% (REFRESH OPTIVE® ADVANCED) administered as 1-2 drops in each eye, as needed, at least 2 times daily for 90 days.
  Interventions: Drug: Carboxymethylcellulose Sodium 0.5%

INTERVENTIONS:
Drug: Carboxymethylcellulose Based Eye Drop — Carboxymethylcellulose based eye drop (OM3 Tear) administered as 1-2 drops in each eye, as needed, at least 2 times daily for 90 days.
  Arms: OM3 Tear
Drug: Carboxymethylcellulose Sodium 0.5% — Carboxymethylcellulose sodium 0.5% (REFRESH OPTIVE® ADVANCED) administered as 1-2 drops in each eye, as needed, at least 2 times daily for 90 days.
  Other Names: REFRESH OPTIVE® ADVANCED
  Arms: REFRESH OPTIVE® ADVANCED

SUMMARY:
This study will evaluate the safety and efficacy of a new eye drop formulation in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Used artificial tears for dry eye
* Visual acuity of at least 20/32 (while wearing glasses, if necessary).

Exclusion Criteria:

* Use of contact lenses in the last 3 months, or anticipated use of contact lenses during the study
* Herpes keratitis in the last 6 months
* Cataract surgery, laser-assisted in situ keratomileusis [LASIK], or photorefractive keratectomy, within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (13):
- United States (10):
  - The Private Practice of Milton Hom, OD, Azusa, California
  - Havana Research Institute LLC, Burbank, California
  - Lugene Eye Institute, Glendale, California
  - Eric M. White, OD, INC, San Diego, California
  - Moyes Eye Center, PC, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Charlotte Eye Ear Nose, Charlotte, North Carolina
  - Scott and Christie and Associate, Cranberry Township, Pennsylvania
  - Texan Eye, Austin, Texas
- Australia (3):
  - Department of Optometry & Vision Sciences, The University of Melbourne, Parkville
  - Prof. M.T. Coroneo Pty. Ltd., Randwick
  - The University of New South Wales School of Optometry and Vision Science, Sydney

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Started | 120 | 122
Completed | 114 | 116
Not Completed | 6 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal of Consent | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other Miscellaneous Reasons | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED | Total
Number analyzed (Participants) | 120 | 122 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (17.3) | 52.8 (16.7) | 53.5 (17.0)
Age, Customized [Number; unit: participants]
  < 30 years | 16 | 14 | 30
  30 to 40 years | 11 | 18 | 29
  > 40 years | 93 | 90 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 95 | 179
  Male | 36 | 27 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Ocular Surface Disease Index© (OSDI©) Score
Description: The OSDI© consists of 12 questions the patient is asked measuring the presence of ocular symptoms. Each of the 12 questions was assessed using a 5-point scale where 0=none of the time and 4=all of the time. The score is converted to a 0 to 100-point score where 0 is no symptoms and 100 is most symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Number analyzed (Participants) | 120 | 122
score on a scale
  Baseline | 41.12 (12.68) | 39.63 (11.33)
  Change at Day 90 | -15.61 (16.52) | -13.16 (17.71)

2. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT)
Description: TBUT is defined as the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. The worse eye is used for the calculations and is defined as the eye with the shortest average TBUT at Baseline. A positive number change from Baseline indicates improvement and a negative number change from Baseline indicates a worsening.
Time Frame: Baseline, Day 90
Population: ITT population included all randomized participants. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Number analyzed (Participants) | 120 | 122
seconds
  Baseline | 4.77 (1.68) | 4.93 (1.74)
  Change at Day 90: number analyzed (Participants) | 115 | 118
  Change at Day 90 | 1.12 (1.93) | 1.34 (2.62)

3. Secondary Outcome: Change From Baseline in Corneal Staining Score
Description: Total corneal staining with fluorescein was measured in the worse eye using a 6-point scale where 0= none, no staining (best) to 5=severe staining (worst). The total score is calculated as the sum of 5 regions of the cornea, resulting in a possible minimum score of 0 and a maximum possible score of 25 (severe staining score of 5 in all 5 regions). The worse eye is defined as the eye with the highest score at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Number analyzed (Participants) | 120 | 122
score on a scale
  Baseline | 4.49 (3.39) | 4.51 (3.29)
  Change at Day 90: number analyzed (Participants) | 115 | 119
  Change at Day 90 | -1.49 (2.37) | -0.58 (2.70)

4. Secondary Outcome: Change From Baseline in Conjunctival Staining Score
Description: Total conjunctival staining with lissamine green was measured in the worse eye using a 6-point scale where 0= none (best), no staining to 5=severe staining (worst). The total score is calculated as the sum of the 6 regions of the conjunctiva, resulting in a minimum possible score of 0 maximum possible score of 30 (severe staining score of 5 in 6 regions). The worse eye is defined as eye with the highest score at Baseline. A negative change from Baseline represents a decrease in staining (improvement).
Time Frame: Baseline, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Number analyzed (Participants) | 120 | 122
score on a scale
  Baseline | 6.73 (5.65) | 5.87 (4.46)
  Change at Day 90: number analyzed (Participants) | 115 | 119
  Change at Day 90 | -1.76 (4.42) | -1.18 (4.03)

5. Secondary Outcome: Change From Baseline in the Schirmer Test
Description: The Schirmer Test measures tears produced by the eye over 5 minutes using a paper strip inserted into the eye. The results indicate the presence of dry eye (Normal = greater than 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye. The worse eye defined as the eye with the lowest score at baseline is used to calculate the change at Day 90. A positive number change from baseline indicates an increase in tears (improvement).
Time Frame: Baseline, Day 90
Population: ITT population included all randomized participants. "n" is the number of participants in the category with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Number analyzed (Participants) | 120 | 122
mm
  Baseline | 9.91 (7.10) | 9.85 (6.82)
  Change at Day 90: number analyzed (Participants) | 115 | 118
  Change at Day 90 | 1.40 (7.13) | 1.38 (7.21)

ADVERSE EVENTS:
Time Frame: 120 Days
Arm/Group | OM3 Tear | REFRESH OPTIVE® ADVANCED
Serious Adverse Events (participants affected / at risk) | 1/120 | 1/122
Other Adverse Events (participants affected / at risk) | 0/120 | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OM3 Tear (N=120) | REFRESH OPTIVE® ADVANCED (N=122)
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.